CLINICAL TRIAL: NCT07187609
Title: Clinical and Radiographic Evaluation of Zinc Incorporated Bovine Derived- Hydroxyappatite Xenograft in Immediately Placed Implant: A Randomized Clinical Study
Brief Title: Zinc Incorporated Bovine Derived- Hydroxyappatite Xenograft in Immediately Placed Implant
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Ibrahim montasser, Resident, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Zinc in immediate implant
Record Dates: First submitted 2025-08-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2024-09

CONDITIONS: Implant; Zinc Status
Keywords: bone grafts; Implant; zinc in corporated bovine drived hydroxyappatite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (control) (Experimental): patients will undergo immediate implant with bovine drived hydroxyapatite xenograft
  Interventions: Procedure: Immediate implant with bovine drived hydroxyapatite xenograft.
- Group II (Test group) (Experimental): patients will undergo immediate implant with zinc incorporated bovine drived hydroxyapatite xenograft
  Interventions: Procedure: immediate implant with zinc incorporated bovine drived hydroxyapatite xenograft

INTERVENTIONS:
Procedure: Immediate implant with bovine drived hydroxyapatite xenograft. — patients will undergo immediate implant with bovine drived hydroxyapatite xenograft.
  Arms: Group I (control)
Procedure: immediate implant with zinc incorporated bovine drived hydroxyapatite xenograft — patients will undergo immediate implant with zinc incorporated bovine drived hydroxyapatite xenograft
  Arms: Group II (Test group)

SUMMARY:
The aim of this study is to evaluate Clinical and radiographic effect of zinc incorporated bovine derived hydroxyapatite xenograft and bovine hydroxyapatite xenograft alone for immediately placed implant

DETAILED DESCRIPTION:
Implant dentistry is a prosthetic effort via a surgical procedure. In order to achieve an ideal prosthetic construct, precise plan should be taken into consideration prior to the beginning of treatment. The position of implant requires protected prosthesis. It can be affected by the implant size, volume, and the quantity and quality of bone provided at various sites.

One pitfall of immediate implant use, however, is the inevitable residual space that remains between the implant body and the socket wall, due to a discrepancy in size between the implant and the socket wall. This space, which is located toward the coronal end of the implant, is called the jumping distance. Excessive jumping distance may lead to bone resorption and formation of a bony defect, decreasing the implant stability .

One of the most extensively used methods for restoration of the lost attachment is the use of bone grafts. bone grafting which is one of the methods used to address these issues has experienced an increased level of demand.

The problem of bone defects has also contributed to making bone autograft become the gold standard for treating bone abnormalities, although it has its limitations which are graft quantity and donor site morbidity. Contributory,allografts have become popular for replacing bone defects because the graft size can be easily adjusted but it also has several drawbacks, including disease transfer, rejection reactions, non-union, graft resorption, fracture, and donor restrictions A xenograft is one of the choices used to overcome these limitations since the raw material is plentiful, readily available, and inexpensive. Additionally, several previous studies showed that organic or inorganic matrix derived from bovine bone is biocompatible, but this biomaterial requires proper preparation to avoid risks such as the transmission of zoonoses .

Bovine hydroxyapatite is made up of materials which have biological properties that makes it biocompatible and osteoconductive. These important biological properties allow the apposition of newly formed bone by osteoprogenitor cells and the partial remodeling by osteoclast and osteoblast of the host . Hydroxyapatite is used as scaffolds to support the development of bone tissue from an osteoblast proliferation stage through to extracellular matrix (ECM) deposition and on to cell-mediated early-stage mineralization. The addition of small quantities of hydroxyapatite to the scaffolds considerably increases calcium deposition and has a mild osteogenic impact.

One of the potential methods for producing anorganic xenograft with enhanced osteoconductivity is by substituting ions with the constituent elements of hydroxyapatite that exist in bone mineral because this method has the potential to increase hydroxyapatite solubility by lowering its crystallinity and inducing a higher number of structural defects. For these reasons, the ionic activity product of apatite increases in body fluid due to the released constituent elements of apatite and this will provoke the formation of low crystalline hydroxyl carbonate apatite (bioactivity) on ions substituted hydroxyapatite surface, which enhances osteoconductivity. However, the effect of other ions in bone on the bioactivity and osteoconductivity of hydroxyapatite has not been extensively investigated. The substitutions of sodium with calcium ions26-38 and chlorine with hydroxyl ions39-50 in hydroxyapatite have been also reported, respectively, but they were confined to synthetic procedures and structural analyses.

Zinc is the most abundant trace metallic element found in the body with 85% present in muscle and bone.Zinc has proven to possess a direct stimulatory effect on osteoblastic cells in vitro while bone resorption was inhibited . It also reduces bacterial load, thus proving its antimicrobial properties. Many studies have demonstrated that zinc significantly improved the bioactivity of HA. Therefore, zinc-HA can be a new generation of materials for bone tissue- engineering.

In comparison with the pure HA group, Zn2+-doped HA had more connective tissues replaced by rebuilt bones, confirming that Zn2+-doped HA had a stronger osteo-induction potential.

In a word, Zn2+ ions act in promoting cell proliferation, increasing osteogenic activity, and inhibiting osteoclast bioactivity. Zn2+-doped HA was considered as a suitable substitute for cancellous bone.

To the best of our knowledge there are no studies conducted on zinc incorporation bovine derived hydroxyapatite xenograft (Zn-BHA) on immediate implant so this study designed to evaluate the effect of bovine drived hydroxyapatite xenograft (BHA) alone and zinc incorporated bovine drived hydroxyapatite xenograft clinically and radographically on immediat implant.

With the advancement of computer-aided design and computer-aided manufacturing (CAD-CAM) technology, there are different approaches for implant prosthetics' digital workflow.

Recent digital technology allowed the virtual extraction of unrestorable teeth, the design of a restoration with a perfect emergence profile that preserves soft tissue contour, and finally the 3D printing of the interim restoration.

The CAD-CAM guided templates have many applications in dentistry such as implant placement and endodontic access preparations, the guided implant osteotomy presents an accurate protocol for implant placement in the preplanned position with less surgical time and few post-surgical complications.

The digitally designed surgical guides transfer the virtually planned implant angulation, width and length through the use of 3D printed transparent template.

ELIGIBILITY:
Inclusion Criteria:

* Adult(male or female) patients between the ages of 21 -50 years who requiring the replacement of one or more non-restorable teeth in the mandible which will be indicated for extraction.
* Adequate bone dimensions at the implant site with ridge width of at least 6 mm, the availability of at least 3mm of sound subapical bone, the presence of an intact labial bone plate, and no evidance of periapical infection on cone beam computed tomography or clinically
* The peri-implant gaps larger than 1.5 mm will be included.
* All patients will be physically healthy with no medical history of any systemic disease.

Exclusion Criteria:

* Smokers.
* Patients with para functional habits such as bruxism and clenching
* Poorly controlled systemic diseases which preclude local anesthesia or surgical procedures
* Patients undergoing chemotherapy or radiotherapy and immuno-compromised patients.
* Pregnant /lactating women.
* Patients that are allergic to zinc
* Patients on antibiotic therapy in the pervious 6 months

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2025-10-08 (Estimated); Study Completion 2026-11-08 (Estimated)

PRIMARY OUTCOMES:
Marginal bone loss | 9 months
  Marginal bone loss was defined as the distance from the implant platform to the alveolar crest.

SECONDARY OUTCOMES:
densitometric gray scale value to measure bone density | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Suez canal university, Suez, Egypt

IPD SHARING:
Plan to Share IPD: No